CLINICAL TRIAL: NCT06464068
Title: AGNOSTIC THERAPY IN A PHASE II, MULTICENTER, SINGLE-ARM STUDY IN FIRST-LINE TREATMENT OF DURVALUMAB IN ASSOCIATION WITH CARBOPLATIN OR CISPLATIN AND ETOPOSIDE IN PATIENTS AFFECTED BY EXTENSIVE STAGE - EXTRAPULMONARY SMALL CELL CARCINOMA
Brief Title: AGNOSTIC THERAPY IN A PHASE II SINGLE-ARM STUDY IN FIRST-LINE TREATMENT OF DURVALUMAB IN ASSOCIATION WITH CARBOPLATIN OR CISPLATIN AND ETOPOSIDE IN PATIENTS AFFECTED BY EXTENSIVE STAGE - EXTRAPULMONARY SMALL CELL CARCINOMA
Acronym: DURVASCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOIRC-01-2021
Record Dates: First submitted 2024-06-07; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Extrapulmonary Small Cell Carcinoma
Keywords: EXTRAPULMONARY SMALL CELL CARCINOMA (EPSCC); DURVALUMAB
MeSH Terms: interventions — durvalumab; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DURVALUMAB IN ASSOCIATION WITH CARBOPLATIN OR CISPLATIN AND ETOPOSIDE (Experimental): All drugs will be administered intravenously. Induction treatment will be administered on a 21-day cycle for four cycles and will consist of:
  * etoposide 80-100 mg/m² (administered on days 1-3 of each 21-day cycle);
  * investigator's choice of either carboplatin area under the curve 5-6 mg/mL per min or cisplatin 75-80 mg/m² (administered on day 1 of each cycle);
  * durvalumab 1500 mg every 3 weeks in combination with chemotherapy (induction phase) followed by maintenance phase with durvalumab 1500 mg every 4 weeks. Patients will continue treatment until disease progression per investigator assessment, unacceptable toxicity, or other discontinuation criteria were met for a maximum of 24 months. Continuation of study treatment after disease progression will be permitted if there is evidence of clinical benefit for a maximum 24 months.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — All drugs will be administered intravenously. Induction treatment will be administered on a 21-day cycle for four cycles and will consist of:
  * etoposide 80-100 mg/m² (administered on days 1-3 of each 21-day cycle);
  * investigator's choice of either carboplatin area under the curve 5-6 mg/mL per min or cisplatin 75-80 mg/m² (administered on day 1 of each cycle);
  * durvalumab 1500 mg every 3 weeks in combination with chemotherapy (induction phase) followed by maintenance phase with durvalumab 1500 mg every 4 weeks. Patients will continue treatment until disease progression per investigator assessment, unacceptable toxicity, or other discontinuation criteria were met for a maximum of 24 months. Continuation of study treatment after disease progression will be permitted if there is evidence of clinical benefit for a maximum 24 months.
  Other Names: Etoposide, Cisplatin. Carboplatin

SUMMARY:
This is a phase II, single-arm, multicenter study to evaluate the activity and safety of durvalumab in combination with carboplatin or cisplatin plus etoposide in patients with treated ES-EPSCC.

DETAILED DESCRIPTION:
All drugs will be administered intravenously. Induction treatment will be administered on a 21-day cycle for four cycles and will consist of:

* etoposide 80-100 mg/m² (administered on days 1-3 of each 21-day cycle);
* investigator's choice of either carboplatin area under the curve 5-6 mg/mL per min or cisplatin 75-80 mg/m² (administered on day 1 of each cycle);
* durvalumab 1500 mg every 3 weeks in combination with chemotherapy (induction phase) followed by maintenance phase with durvalumab 1500 mg every 4 weeks. Patients will continue treatment until disease progression per investigator assessment, unacceptable toxicity, or other discontinuation criteria were met for a maximum of 24 months. Continuation of study treatment after disease progression will be permitted if there is evidence of clinical benefit for a maximum 24 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years on day of signing informed consent. 2. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.

  3. Histologically or cytologically confirmed extensive disease extrapulmonary small cell carcinoma.

  4. Brain metastases; must be asymptomatic or treated and stable off steroids and anti-convulsant for at least 1 month prior to study treatment. Patients with suspected brain metastases at screening should have a CT/MRI of the brain prior to study entry. 5. No prior exposure to immune-mediated therapy, including durvalumab excluding therapeutic anticancer vaccines. 6. No prior exposure to chemotherapy for advance disease. 7. Performance status of 0 or 1 on the ECOG Performance Scale. 8. Life expectancy ≥12 weeks at enrollment (day 1). 9. Patients must be considered suitable to receive a platinum-based chemotherapy regimen as first-line treatment for ES-EPSCC. 10. Adequate organ and marrow function, all screening labs should be performed within 14 days of treatment initiation:
  1. Haemoglobin ≥9.0 g/dL
  2. Absolute neutrophil count (ANC) ≥1.0 × 109 /L
  3. Platelet count ≥75 × 109/L
  4. Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). <<This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.>>
  5. AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which
  6. case it must be ≤5x ULN 11. Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft- Gault formula. 12. Availability of an archived tumor tissue block at baseline. 13. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female premenopausal patients. 14. At least 1 lesion, not previously irradiated, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes, which must have a short axis ≥15 mm) with CT o MRI, suitable for repeated measurements as per RECIST 1.1 criteria. 15. Body weight >30 kg

     Exclusion Criteria:
* Subjects with active, known or suspected autoimmune disease requiring systemic treatment (systemic steroids or immunosuppressive agents) prior 14 days before the first dose of durvalumab.

The following are exceptions to this criterion:

* Intranasal, inhaled, topical steroids or local steroid injections (eg, intra articular injection).
* Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
* Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
* Premedication with steroids for chemotherapy is acceptable
* Additional malignancy in the last 5 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Any concurrent chemotherapy, investigational product, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable.
* Any history of radiotherapy prior to systemic therapy. Radiation therapy for palliative care (ie, bone metastasis) is allowed but must be completed before first dose of the study medication.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis with the exception of diverticulosis, systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, and uveitis, etc]).

The following are exceptions to this criterion:

* Patients with vitiligo or alopecia
* Patients with hypothyroidism (eg, following Hashimoto syndrome) and stable on hormone replacement
* Any chronic skin condition that does not require systemic therapy
* Patients without active disease in the last 5 years may be included but only after consultation with the Study Physician
* Patients with celiac disease controlled by diet alone

  * Major surgical procedure within 28 days prior to the first dose of investigational product. Local surgery of isolated lesions for palliative intent is acceptable.
  * History of leptomeningeal carcinomatosis.
  * History of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
  * Active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
  * Receipt of live, attenuated vaccine within 30 days prior to the first dose of investigational product.

Patients, if enrolled, should not receive live vaccine whilst receiving the investigational product and up to 30 days after the last dose of investigational product.

* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* History of allogenic organ transplantation.
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart)
* Female patients with a positive pregnancy test at enrollment or prior to administration of study medication
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy (for more information, refer to paragraph 10.8) .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
progression free survival (PFS) | 12 months
  To evaluate the preliminary efficacy in terms of 12 months progression free survival (PFS) of durvalumab in association with carboplatin or cisplatin and etoposide in first line patients affected by extensive stage EPSCC. PFS isdefined as the time from initiation of study treatment to the first occurrence of disease progression or death from any cause, whichever occurs first. According to the results of the CASPIAN trial [18] in which was observed a 12-month progression-free survival rates of 5% (2.4-8.0) for patients that had received Platinum-etoposide, it is expected to detect an increasing of at least 10 percentage points (to 15%).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 12 months
  Activity of durvalumab in combination with carboplatin or cisplatin plus etoposide in patients with untreated extensive- stage extrapulmonary small cell lung cancer (EPSCC). Activity will be measured as Objective Response Rate (ORR), defined as the percentage of patients who attain complete response (CR) or partial response (PR) according to RECIST v1.1.
Disease control rate (DCR) | 12 months
  Disease control rate (DCR) measured as the percentage of patientswho have archived CR, PR, and stable disease (SD).
Overall survival (OS) | 24 months
  Overall survival (OS), defined as the time from initiation of study treatment to death from any cause.
Duration of response (DOR) | 12 months
  Duration of response (DOR), is defined as the time from initial response to disease progression or death among patients who have experienced a CR or PR (unconfirmed) during the study. Duration of response will be calculated based on disease status evaluated by the investigator according to RECIST v1.1.
quality of life (QoL) | 24 months
  To describe change in quality of life of patients during the study, measured as pre-defined PRO endpoints in this study are mean change from baseline in questionnaire administred at the enrollment time (baseline) and after the induction phase (3 +/- 2 weeks)
incidence, nature, frequency, and severity of Adverse Events (AEs) | 24 months
  Safety profile of durvalumab, defined in terms of incidence, nature, frequency, and severity of Adverse Events (AEs) and laboratory abnormalities graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0;

OTHER OUTCOMES:
biomarkers associated with sensitivity/resistance to immune checkpoint inhibitors | 24 months
  To identify possible biomarkers associated with sensitivity/resistance to immune checkpoint inhibitors, tumor samples from enrolled patients will undergo whole exome sequencing (WES) and gene expression profiling by using a 3' RNA Seq approach.
  For all the patients enrolled to investigate the occurrence of genetic alterations that might be associated with acquired resistance to immune checkpoint inhibitors, blood samples will be collected by analyzing the circulating free DNA (cfDNA). To this end, plasma will be collected at baseline, prior to cycle 5, and at the end of treatment (progression of disease). The cfDNA will be analyzed by targeted sequencing panels.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Damato, MD, Principal Investigator — AUSL/IRCCS of Reggio Emilia
Locations (1):
- AUSL-IRCCS of Reggio Emilia, Reggio Emilia, Italy

REFERENCES:
- [Derived] Damato A, Maglietta G, Antonuzzo L, Berardi R, Buonadonna A, Brighi N, Cinieri S, Di Micco C, Gelsomino F, Grossi F, Martinelli E, Cesario S, Pusceddu S, Spada F, Iachetta F, Gervasi E, Ciardiello G, Normanno N, Pinto C. Agnostic phase II, multicenter, single-arm study with DURVAlumab plus carboplatin or cisplatin and etoposide as first-line treatment in extensive stage - Extrapulmonary Small Cell Carcinoma (EPSCC) patients - DURVASCC trial (GOIRC-01-2021). BMC Cancer. 2025 Nov 12;25(1):1763. doi: 10.1186/s12885-025-15112-w. PMID 41225446